CLINICAL TRIAL: NCT02735187
Title: Monocenter, Randomized, Blinded, Intraindividual Study Evaluating Efficacy and Safety of Blue Light (453 nm) Treatment for Mild Psoriasis Vulgaris Over Three Months Compared to Vitamin D
Brief Title: Efficacy and Safety of Blue Light (453 nm) Treatment for Mild Psoriasis Vulgaris Over Three Months Compared to Vitamin D.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Electronics Nederland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Psoriasis-CT03
Record Dates: First submitted 2016-03-16; First posted 2016-04-12 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- group30 (Active Comparator): Treatment of the target area with 30 minutes of blue light at 453nm compared to Vitamin D creme Daivonex on contralateral Plaque of same patient.
  Interventions: Device: Blue light treatment; Drug: Vitamin D
- group15 (Active Comparator): Treatment of the target area with 15 minutes of blue light at 453nm compared to Vitamin D creme Daivonex on contralateral Plaque of same patient.
  Interventions: Device: Blue light treatment; Drug: Vitamin D

INTERVENTIONS:
Device: Blue light treatment — Phototherapy of localized psoriasis vulgaris plaque with a wearable device emitting blue light at 453nm.
Drug: Vitamin D — Treatment of contralateral localized psoriasis vulgaris plaque with Vitamin D creme (Daivonex)

SUMMARY:
Patients will be screened up to 28 days before start of treatment. During the screening visit, the purpose and procedures of the study will be explained to potential patients and informed consent will be obtained.

At the baseline visit, all inclusion and exclusion criteria will be re-assessed. Eligible patients will be randomized to treatment of the target area with either 30 minutes (group30) or 15 minutes (group15) blue light at 600 milliwatt per square centimeter (mW/cm²). Additionally, two study areas with similar clinical symptomatology will be determined and will be randomized to blue light treated area and Daivonex (Vitamin D) treated area.

After randomization, patients will be trained on a demonstrator device (no actual treatment to ensure investigator is blinded as to which group the patient is randomized to) as well as the Daivonex cream. After patients have been instructed, treatment of the areas will be applied daily (once per day, 5-7 times / week) at home for a treatment period of 12 weeks. During those 12 weeks, patients will return to the study site for safety and effectiveness assessments at week 2, 4, 8 and week 12. A phone call visit will be performed after one week of treatment to check for any adverse events or problems in handling the device or the cream. The visit at week 12 serves as end of treatment visit. The patients will be followed-up for another 4 weeks. Treatment responses will be photo documented.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent prior to any study-mandated procedure
2. Good health as determined by the Investigator
3. Willing and able to comply with study requirements
4. Skin type I-IV according to Fitzpatrick
5. Mild plaque-type psoriasis vulgaris with a Psoriasis Area and Severity Index (PASI) ≤ 10 and body surface area (BSA) ≤ 10 at screening.
6. Presence of two comparable psoriatic plaques suitable to be defined as study areas as follows:

   * located on extremities (plaques located on the palms or sole of the feet are not suitable)
   * Both areas located either on lower or upper extremity
   * Can be located on the same extremity
   * Distance between the two study areas ≥ 11cm (border to border)
   * If lesion is too large to be fully covered, partial treatment possible
7. Otherwise healthy according to physical examination
8. Aged 18 years up to ≤74 years
9. Reliable method of contraception for women of childbearing potential (i.e. low failure rate less than 1per cent per year; e.g. oral contraceptives, intra-uterine device (IUD) or transdermal contraceptive patch)
10. Willing to abstain from excessive sun / UV exposure (e.g. sunbath, solarium) during the course of the study

Exclusion Criteria:

General

1. Inmates of psychiatric wards, prisons, or other state institutions
2. Investigator or any other team member involved directly or indirectly in the conduct of the clinical study
3. Participation in another clinical trial within the last 30 days
4. Pregnant or lactating women Medical History
5. Photodermatosis and/or Photosensitivity
6. Porphyria and/or hypersensitivity to porphyrins
7. Patients with current diagnosis of erythrodermic, exfoliative or pustular psoriasis
8. Congenital or acquired immunodeficiency
9. Patients with any of the following conditions present on the study areas: naevi or signs of hyperpigmentation, viral (e.g. herpes or varicella) lesions of the skin, fungal and bacterial skin infections, parasitic infections and atrophic skin
10. Patients with any of the following conditions present or who have been diagnosed in the past with any of the following conditions on the study areas: skin cancer, severe actinic damage and other precancerous lesions
11. Patients with genetic deficiencies attached with increased sensitivity to light or increased risk to dermatologic cancer ( i.e. Xeroderma pigmentosum, Cockayne Syndrome, Bloom-Syndrome) Concomitant medication/treatment in medical history and during the study Required

    * Treatment of target and control area with Excipial U10 Lipolotio (Galderma)
    * Treatment of control area with Daivonex (Leo Pharma) Allowed
    * Topical treatment of non-study areas with Vitamin D or WHO group I-II corticosteroids or mometasone Not allowed Within 3 months prior to baseline
    * ustekinumab Within 2 months prior to baseline
    * adalimumab, alefacept, infliximab Within 1 month prior to baseline
    * Etanercept
    * Systemic corticosteroids
    * Retinoids
    * Immunosuppressants (e.g. methotrexate, ciclosporin, azathioprine, chemotherapeutics)
    * oral psoralen with ultraviolet A (PUVA)
    * Topical or intranasal/inhalation therapy with potent or very potent (WHO group III-IV) corticosteroids

Within 2 weeks prior to baseline

* ultraviolet B light (UVB) / ultraviolet A light (UVA)
* Topical therapy with
* WHO group I-II corticosteroids
* Topical retinoids
* Vitamin D analogues
* Topical immunomodulators (e.g. calcineurin inhibitors)
* Anthracen derivatives
* Tar
* Salicylic acid
* Intranasal/inhalation therapy with WHO group I-II corticosteroids At baseline

  * Photo-sensitizing medication (e.g. psoralen, tetracycline, nalidixic acid, furosemide, amiodarone, phenotiacine, chinclone, fibrates, hypericumperforatum, arnica, valerian, tar, psoralen, ketoprofen) or colours (e.g. thiazide, toluidine blue, eosin, methylene blue, rose Bengal, acridine)
  * Initiation of, or expected changes in concomitant medication that may affect psoriasis vulgaris (e.g., beta blockers, anti-malaria drugs, lithium and angiotensin converting enzyme (ACE) inhibitors)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Verena von Felbert, PD Dr., Principal Investigator — Universityclinic of the RWTH Aachen
Locations (1):
- Department of Dermatology and Allergology, Medical faculty of the RWTH Aachen, Aachen, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total number of 51 patients were enrolled for the study at 1 study site in Germany between March and April 2016. 140 patients were pre-screened.
Groups:
- group30: Treatment of the target area with 30 minutes of blue light at 453nm compared to VitaminD creme Daivonex on contralateral Plaque of same patient.
  Blue light treatment: Phototherapy of localized psoriasis vulgaris plaque with a wearable device emitting blue light at 453nm.
  Vitamin D: Treatment of contralateral localized psoriasis vulgaris plaque with Vitamin D creme (Daivonex)
- group15: Treatment of the target area with 15 minutes of blue light at 453nm compared to VitaminD creme Daivonex on contralateral Plaque of same patient.
  Blue light treatment: Phototherapy of localized psoriasis vulgaris plaque with a wearable device emitting blue light at 453nm.
  Vitamin D: Treatment of contralateral localized psoriasis vulgaris plaque with Vitamin D creme (Daivonex)
Period: Overall Study
Arm/Group | group30 | group15
Started | 25 | 26
Completed | 21 | 25
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | group30 | group15 | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (13.4) | 47.9 (13.7) | 45.2 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 12 | 10 | 22
Region of Enrollment [Number; unit: participants]
  Germany | 25 | 26 | 51
Skin type [Count of Participants; unit: Participants] — Skin type was assessed by a dermatologist according to Fitzpatrick type (I-VI):
  Type I always burns, never tans (pale white; blond or red hair; blue eyes; freckles).
  Type II usually burns, tans minimally (white; fair; blond or red hair; blue, green, or hazel eyes) Type III sometimes mild burn, tans uniformly (cream white; fair with any hair or eye color) Type IV burns minimally, always tans well (moderate brown) Type V very rarely burns, tans very easily (dark brown) Type VI Never burns, never tans (deeply pigmented dark brown to darkest brown)
  Participants
    Type I | 1 | 0 | 1
    Type II | 12 | 17 | 29
    Type III | 12 | 9 | 21
    Type IV | 0 | 0 | 0
    Type V | 0 | 0 | 0
    Type VI | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Visit 2) of the Local PSI of the Blue Light Treated Area (Group 30) as Compared to the VitaminD Treated Area (Control) at End of Treatment (Week 12).
Description: The local Psoriasis severity index (LPSI) was adapted from the well known PASI. The investigator evaluated and graded the severity of erythema, induration, and scaliness as the key symptoms of psoriasis on the study areas (0-4). A total severity score was calculated as the sum of the three symptom ratings (range 0-12). The measure reported is the change in LPSI at end of treatment versus baseline. A negative change indicates an improvement of the LPSI.
Time Frame: week 12
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- group30 (Blue Light): Treatment of the target area with 30 minutes of blue light at 453nm
- group30 (Comparator): Vitamin D: Treatment of contralateral localized psoriasis vulgaris plaque with Vitamin D creme (Daivonex)
Arm/Group | group30 (Blue Light) | group30 (Comparator)
Number analyzed (Participants) | 25 | 25
units on a scale | -2.4 (1.45) | -2.4 (1.38)
Statistical Analysis 1: Comparison: group30 (Blue Light) vs group30 (Comparator); Test type: Superiority — A paired t-test was applied to test the primary hypothesis. In case the requirements for normality were not met, a non-parametric analysis (Wilcoxon signed rank test) was performed; p = 0.6469, t-test, 2 sided — A probability (P-Value) above 0.05 is considered not to be statistical significant

2. Secondary Outcome: Change From Baseline (Visit 2) of the Local PSI of the Blue Light Treated Area (Group 15) as Compared to the VitaminD Treated (Control) Area at End of Treatment (Week 12).
Description: The local Psoriasis severity index (LPSI) was adapted from the well known PASI. The investigator evaluated and graded the severity of erythema, induration, and scaliness as the key symptoms of psoriasis on the study areas (0-4 each). A total severity score was calculated as the sum of the three symptom ratings (range 0-12). The measure reported is the change in LPSI at end of treatment versus baseline. A negative change indicates an improvement of the LPSI.
Time Frame: week 12
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- group15 (Blue Light): Treatment of the target area with 30 minutes of blue light at 453nm
- group15 (Comparator): Vitamin D: Treatment of contralateral localized psoriasis vulgaris plaque with Vitamin D creme (Daivonex)
Arm/Group | group15 (Blue Light) | group15 (Comparator)
Number analyzed (Participants) | 26 | 26
units on a scale | -2.4 (1.65) | -2.5 (1.56)

3. Secondary Outcome: Change From Baseline in Patient Self-assessment of Severity of Psoriasis of the Blue Light Treated Area (Group 30) Compared to the VitaminD Treated (Control) Area at Week 12 (VAS Scale).
Description: Patient Rating of severity of Psoriasis Plaques on a 0-10 cm Visual Analogue Scale (VAS) scale. VAS = 0 cm corresponds to no pain,, VAS = 10 cm corresponds to maximal imaginable pain.
Time Frame: week 12
Population: Full Analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | group30 (Blue Light) | group30 (Comparator)
Number analyzed (Participants) | 25 | 25
units on a scale | -3.82 (2.70) | -3.56 (2.73)

4. Secondary Outcome: Change From Baseline in Patient Self-assessment of Severity of Psoriasis of the Blue Light Treated Area (Group 15) Compared to the VitaminD Treated (Control) Area at Week 12 (VAS Scale).
Description: Patient Rating of severity of Psoriasis Plaques on 0-10 cm Visual Analogue Scale (VAS) scale. VAS = 0 corresponds to no symptoms of Psoriasis, VAS = 10 corresponds to most severe symptoms of Psoriasis.
Time Frame: week 12
Population: Full Analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | group15 (Blue Light) | group15 (Comparator)
Number analyzed (Participants) | 26 | 26
units on a scale | -2.92 (2.44) | -2.44 (2.79)

5. Secondary Outcome: Lesional Erythema Measured by Mexameter Measured at End of Treatment.
Description: Lesional erythema was measured objectively with a measurement device (Mexameter). The Mexameter delivers a two digit number for the redness of the skin (range 0-99). 0 = no redness and 99 = maximal redness.
Time Frame: week 12
Population: Full Analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- group15 (Blue Light): Treatment of the target area with 15 minutes of blue light at 453nm
Arm/Group | group30 (Blue Light) | group30 (Comparator) | group15 (Blue Light) | group15 (Comparator)
Number analyzed (Participants) | 25 | 25 | 26 | 26
units on a scale | 65.44 (16.29) | 65.32 (14.27) | 59.88 (10.94) | 61.50 (11.75)

6. Secondary Outcome: Patient Satisfaction (Week 12)
Description: Patient satisfaction will be measured by questionnaire using the System usability score (SUS). The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. Though the scores are 0-100, these are not percentages and should be considered only in terms of their percentile ranking. The higher the score the better the patient satisfaction the better the outcome. The lower the score the worse the patient satisfaction the worse the outcome.
Time Frame: week 12
Population: Full Analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | group30 | group15
Number analyzed (Participants) | 21 | 20
units on a scale | 88.62 (7.92) | 89.00 (8.71)

7. Other Pre Specified Outcome: Hyperpigmentation of Treated Skin Areas Exposed to Blue Light and Control Area Exposed to Daivonex- Evaluation by Mexameter
Description: Lesional tanning was measured objectively with a measurement device (Mexameter). The Mexameter delivers a two digit number for the brownish color of the skin (range 0-99). 0 = no tanning and 99 = maximal tanning.
Time Frame: week 2-16
Population: Safety Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | group30 (Blue Light) | group30 (Comparator) | group15 (Blue Light) | group15 (Comparator)
Number analyzed (Participants) | 25 | 25 | 26 | 26
units on a scale
  week 2 | 26.72 (7.20) | 24.16 (3.77) | 24.65 (6.72) | 22.92 (3.78)
  week 4 | 25.48 (5.95) | 24.52 (5.93) | 24.15 (3.90) | 23.12 (3.60)
  week 8 | 27.40 (6.89) | 25.00 (4.21) | 25.31 (8.99) | 22.35 (6.24)
  week 12/End of treatment | 25.60 (5.11) | 24.96 (4.23) | 26.15 (5.90) | 24.15 (5.96)
  week 16 | 25.76 (4.61) | 25.16 (4.67) | 26.31 (7.04) | 25.04 (7.13)

8. Other Pre Specified Outcome: Adverse Events (Serious and Non-serious)
Description: Adverse Events (serious and non-serious) collected during the study conduct.
Time Frame: week 0-16
Population: Safety set
Measure: Number; unit: Number of adverse events
Arm/Group | group30 | group15
Number analyzed (Participants) | 25 | 26
Number of adverse events
  Any adverse events | 4 | 10
  Causal related to IMD | 0 | 0
  Causal related to medical procedure | 1 | 0

9. Other Pre Specified Outcome: Adverse Device Effects
Description: Adverse device effects collected during the study conduct.
Time Frame: week 0-16
Population: Safety set
Measure: Number; unit: Number of adverse device effects
Arm/Group | group30 | group15
Number analyzed (Participants) | 25 | 26
Number of adverse device effects | 0 | 0

10. Other Pre Specified Outcome: Device Deficiencies
Description: The number of device deficiencies was collected throughout the study
Time Frame: week 0-12
Population: Safety set
Measure: Number; unit: Number of device deficiencies
Arm/Group | group30 | group15
Number analyzed (Participants) | 25 | 26
Number of device deficiencies | 2 | 2

11. Other Pre Specified Outcome: Thermal Comfort
Description: Thermal comfort will be measured by questionaire: How comfortable was this temperature on your skin?
Time Frame: week 12
Population: Safety set
Measure: Number; unit: Count of Participants
Arm/Group | group30 | group15
Number analyzed (Participants) | 25 | 26
Count of Participants
  Very uncomfortable | 0 | 0
  Uncomfortable | 0 | 0
  Slightly uncomfortable | 5 | 4
  Just right | 9 | 8
  Slightly comfortable | 2 | 3
  Comfortable | 7 | 10
  Very comfortable | 0 | 0
  No data | 2 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the complete 16 weeks of the clinical Investigation.
Description: Any untoward medical occurrence, unintended disease or injury, or any untoward clinical signs (including an abnormal laboratory finding) in patients, users or other persons whether or not related to the investigational medical device. This includes events related to the investigational device or the comparator. This includes events related to the procedures involved. For users or other persons this is restricted to events related to the investigational medical device.
Arm/Group | group30 | group15
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/25 | 3/26
Other Adverse Events (participants affected / at risk) | 4/25 | 10/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | group30 (N=25) | group15 (N=26)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Not related to investigational medical device (IMD) or medical procedure
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Not on investigational site, not related to IMD or medical procedure
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1) — Not related to IMD or medical procedure
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | group30 (N=25) | group15 (N=26)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Endoscopy upper gastrointestinal tract (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No